CLINICAL TRIAL: NCT01737879
Title: Evaluation of the Conversion From Peginesatide to Epoetin Alfa in Subjects Receiving Hemodialysis
Brief Title: Evaluation of the Conversion From Peginesatide to Epoetin Alfa in Patients Receiving Hemodialysis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated: Test article, Omontys, was recalled from the market; Enrollment has halted prematurely and will not resume; participants are no longer being treated
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110209
Record Dates: First submitted 2012-10-03; First posted 2012-11-30 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Anemia
Keywords: Anemia, Chronic Kidney Disease, End Stage Renal Disease, erythropoiesis-stimulating agents, Hemodialysis, Hemoglobin
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — peginesatide; hematide; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginesatide / Epoetin Alfa (Experimental): Participants were treated with peginesatide administered intravenously (IV) every 4 weeks for 24 weeks. Participants were then to be converted back to epoetin alfa administered by IV 3 times a week for 32 weeks.
  Interventions: Drug: Peginesatide; Drug: Epoetin alfa

INTERVENTIONS:
Drug: Peginesatide — All participants will receive peginesatide for the first 24 weeks.
  Other Names: Omontys
Drug: Epoetin alfa — All participants converted to epoetin alfa at week 25 for a total of 32 weeks
  Other Names: Epogen

SUMMARY:
The purpose of this study is to evaluate whether hemodialysis patients on peginesatide can be converted to epoetin alfa by using a predefined conversion table while achieving a stable hemoglobin.

DETAILED DESCRIPTION:
This is a phase 4, multicenter, single-arm, open-label study designed to evaluate whether patients receiving hemodialysis and treated with peginesatide can be converted to epoetin alfa using a predefined conversion table while achieving stable hemoglobin. The study will be conducted in two phases. Hemodialysis patients treated with epoetin alfa 3 times a week (TIW) will first be converted to peginesatide administered every 4 weeks (Q4W). After 24 weeks, these participants will be converted back to epoetin alfa administered TIW for 32 weeks. The primary endpoint will be the mean hemoglobin during the last 8 weeks of the epoetin alfa period.

ELIGIBILITY:
Key Inclusion Criteria:

* Receiving hemodialysis 3 times a week
* Receiving epoetin alfa IV 3 times a week
* Hemoglobin concentration ≥ 9.0 and ≤ 12.0 g/dL within 8 weeks of or during screening

Key Exclusion Criteria:

* Systemic hematologic disease
* Changes in Epoetin alfa dose by ≥ 50% within 8 weeks of or during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (23):
- United States (23):
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Azusa, California
  - Research Site, Bakersfield, California
  - Research Site, Granada Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Paramount, California
  - Research Site, Riverside, California
  - Research Site, Whittier, California
  - Research Site, Orange, Connecticut
  - Research Site, Meridian, Idaho
  - Research Site, Kansas City, Missouri
  - Research Site, Bayonne, New Jersey
  - Research Site, Amherst, New York
  - Research Site, Yonkers, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Orangeburg, South Carolina
  - Research Site, Dyersburg, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Chesapeake, Virginia

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled on 24 October 2012; Last patient was enrolled on 21 February 2013. The study was terminated on 27 March 2013.
Groups:
- Peginesatide: Participants were treated with peginesatide administered intravenously (IV) every 4 weeks for 24 weeks. Participants were then to be converted back to epoetin alfa administered by IV 3 times a week for 32 weeks.
Period: Overall Study
Arm/Group | Peginesatide
Started | 41
Received Peginesatide | 34
Transitioned to Epoetin Alfa | 0
Completed | 0
Not Completed | 41
Not completed — Death | 1
Not completed — Sponsor decision | 40

BASELINE CHARACTERISTICS:
Arm/Group | Peginesatide
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 24
  White | 16
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Hemoglobin Concentration During the Evaluation Period
Description: The hemoglobin concentrations during the evaluation period after the conversion to epoetin alfa were to be averaged for each participant and then summarized over all participants.
  No participant reached the evaluation period, therefore, the primary efficacy endpoint could not be evaluated.
Time Frame: Last 8 weeks of epoetin alfa treatment period period (Weeks 49 to 56).
Arm/Group | Peginesatide
Number analyzed (Participants) | 0

2. Secondary Outcome: Mean Dose of Epoetin Alfa During the Evaluation Period
Description: No participant reached the evaluation period, therefore, this endpoint could not be evaluated.
Time Frame: Last 8 weeks of epoetin alfa treatment period period (Weeks 49 to 56).
Arm/Group | Peginesatide
Number analyzed (Participants) | 0

3. Secondary Outcome: Hemoglobin Concentration by Visit
Time Frame: Baseline and Weeks 3, 5, 7, 9, 11, 13, 15, 17, 19, and 21
Population: Primary analysis set includes all enrolled participants who received at least 1 dose of investigational product. The number of participants with available data at each time point is indicated by "n".
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide
Number analyzed (Participants) | 34
g/dL
  Baseline (n=34) | 10.51 (0.76)
  Week 3 (n=34) | 11.09 (0.81)
  Week 5 (n=29) | 10.86 (0.87)
  Week 7 (n=21) | 11.03 (1.02)
  Week 9 (n=20) | 10.59 (0.84)
  Week 11 (n=19) | 10.80 (0.97)
  Week 13 (n=14) | 10.50 (0.94)
  Week 15 (n=10) | 10.70 (0.82)
  Week 17 (n=10) | 10.35 (1.31)
  Week 19 (n=10) | 10.93 (0.94)
  Week 21 (n=1) | 10.10 (NA) — Data only available for one participant
  End of study visit (n=32) | 10.55 (0.63)

4. Secondary Outcome: Peginesatide Dose by Visit
Time Frame: Baseline and Weeks 5, 9, 13, and 17
Population: Primary analysis set, with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Peginesatide
Number analyzed (Participants) | 34
mg
  Baseline (n=30) | 5.42 (2.48)
  Week 5 (n=16) | 5.04 (1.32)
  Week 9 (n=15) | 4.98 (2.00)
  Week 13 (n=9) | 4.00 (2.53)
  Week 17 (n=9) | 5.12 (3.29)

ADVERSE EVENTS:
Time Frame: From informed consent up to 30 days post treatment, or end of study. Maximum time on study was 6 months.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Peginesatide
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 6/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=34)
Ventricular asystole (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=34)
Oedema (General disorders) | 2
Headache (Nervous system disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.